CLINICAL TRIAL: NCT05216874
Title: The Effect of Splint Usage in Laterognathic Cl III Orthognathic Surgery Patients: Controlled Clinical Trial
Brief Title: The Effect of Splint Usage in Laterognathic Cl III Orthognathic Surgery Patients
Acronym: TMJ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Banu Kılıç, Assistant Professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: laterognathia MPI
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Skeletal Malocclusion; Class III Malocclusion; Laterognathia
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Intervention Model Description: Preoperative occlusal splint treatment Cl III Laterognathia patients
Who Masked: Participant
Masking Description: Although it will be explained to the patients that they would be included in a study determining the joint positions and that a bite record would be taken from them during the operation for this purpose, they will not informed about whether they are included in the splint treatment group or the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusal stabilization splint (Experimental): Skeletal class III laterognathia surgery patients who has occlusal stabilization splint thearapy for at least 2 mounths before surgery
  Interventions: Device: Oclusal Splint
- Control (No Intervention): Skeletal class III laterognathia surgery patients did not have occlusal stabilization splint thearapy

INTERVENTIONS:
Device: Oclusal Splint — Cl III Laterognati volunteer group using occlusal stabilization splint before orthognathic surgery
  -Splint will be used for at least two months
  Arms: Occlusal stabilization splint

SUMMARY:
It is crucial to maintain the anatomic condylar positions during orthognathic surgery. Condylar positions are affected directly under general anesthesia because of joint and muscle relaxation. Possible unwanted changes in the joint position may cause incorrect positioning of the jawbones. This could affect the success of the surgery in terms of function and facial aesthetics causing the need for a second surgery. Our aim is to evaluate whether the use of MR Splint has a statistically significant effect on muscle relaxation-induced condyle position deviations under general anesthesia in Class III Laterognathia patients.

DETAILED DESCRIPTION:
It is crucial to maintain the anatomic condyle positions during orthognathic surgery to prevent iatrogenic temporomandibular joint complications. Condyle shunts are affected directly under general anesthesia because of the joint and muscle relaxation. Surgical guidance appliances are prepared according to the TMJ records taken chairside while patients are in an upright position. During surgery, these appliances are applied in a supine position while the muscles are relaxed. Postoperative and long-term effects of TMJ and muscle relaxation obtained under general anesthesia in class III and asymmetric patients will be examined. Patients who had occlusal splint before records taken will be evaluated in terms of condyle location by MPI.

Our aim is to evaluate whether the use of MR Splint has a statistically significant effect on muscle relaxation-induced condyle position deviations under general anesthesia in Class III Laterognathia patients.

ELIGIBILITY:
Inclusion Criteria:

* being ready for orthognathic surgery
* must be able to give centric relation records

Exclusion Criteria:

* having any TMDsyndromes
* cleft lip and palate,
* have bruxism,
* TMJ or muscle disfunctions,
* under any medication of muscle relaxants,
* narcotics and antidepressants,
* usage of removeable prosthetics
* have toothless areas that can affect the wax impression for centric record
* used horizontal elastics within the last 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-08-20 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
MPI Records for Splint Users | 12 months
  Difference between preoperative and intraoperative condylar positions will be observed as mm with bite records. MPI will be used in the lab to determine the difference.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kılıç, asst. prof, Study Director — Bezmialem Vakıf Üniversitesi
Locations (1):
- Banu Kılıç, Fatih, Istanbul, Turkey (Türkiye)